CLINICAL TRIAL: NCT05363553
Title: Transition to Infant Formula Feeding on Gastrointestinal Regurgitation (TIGER) Study
Acronym: TIGER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dairy Goat Co-operative (N.Z.) Limited (Industry)
Collaborators: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DGC202106
Record Dates: First submitted 2022-04-21; First posted 2022-05-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Gastrointestinal Disorder, Functional; Regurgitation, Gastric; Colic, Infantile; Constipation - Functional; Infant Development
Keywords: infant formula; goat milk; regurgitation
MeSH Terms: conditions — Gastrointestinal Diseases; Laryngopharyngeal Reflux; Colic; Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadrupole
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- infant formula based on whole goat milk (Experimental)
  Interventions: Dietary Supplement: Infant formula based on whole goat milk
- Infant formula based on cow milk proteins (Active Comparator)
  Interventions: Dietary Supplement: infant formula based on cow milk proteins
- Predominantly breastmilk (No Intervention)

INTERVENTIONS:
Dietary Supplement: Infant formula based on whole goat milk — Infant formula based on whole goat milk, nutritionally suitable for infants aged 0-6 months
  Arms: infant formula based on whole goat milk
Dietary Supplement: infant formula based on cow milk proteins — Infant formula based on cow milk proteins, nutritionally suitable for infants aged 0-6 months
  Arms: Infant formula based on cow milk proteins

SUMMARY:
To compare the frequency of regurgitation and other digestive outcomes between infants who receive an infant formula based on whole goat milk and an infant formula based on cow milk proteins during the transition period from breastfeeding to formula feeding, using predominantly breastfed infants as a reference group.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, parallel-group trial to study the effect of feeding infants goat milk or cow milk formula in the first 6 months of life on the prevalence of functional gastrointestinal disorders and other health outcomes, including gastrointestinal health and sleep during the transition from breastfeeding to formula-feeding. A predominantly breastfed group is used as a reference group.

ELIGIBILITY:
Inclusion Criteria:

* healthy full-term born infants (≥ 37 weeks + 0 days and < 41 weeks + 6 days of gestation)
* birth weight ≥ 2.5 kg and ≤ 4.5 kg
* born from a singleton pregnancy
* live in Bangkok or nearby with no plan for geographical migration before 6 months of age
* for experimental and active comparator groups only: parent(s) has expressed the intention to partially (in combination with breastfeeding) or fully formula-feed the infant and ready to enroll in the study before the age of 4 months/120 days
* for no intervention group only: parent(s) has expressed the intention to predominantly breastfeed (according to study definition) and ready to enroll in the study before the age of 4 months/120 days
* infant has been predominantly breastfed for at least 2 weeks before enrollment
* parent(s) has sufficient Thai language skills to understand the study information, the informed consent, and to comply with the study procedure
* parent(s) is willing and deemed able to fulfil the requirements of the study protocol and procedures
* at least one parent is of legal age of consent

Exclusion Criteria:

* infant has any disorder considered to interfere with nutrition, growth or development of the immune system
* participation of the infant in any other interventional trial or participation of the mother in any intervention trial with infant follow-up
* for experimental and active comparator groups only: infant has been formula-fed for more than 1 week before enrolment
* for experimental and active comparator groups only: cow milk allergy or intolerance of the infant
* for experimental and active comparator groups only: enrolled infant who never consumed any study product until the first visit 2 weeks following enrolment

Ages: 2 Weeks to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 146 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Change in daily frequency of regurgitation during the transition period from breastfeeding to formula feeding | From Day 0 to Day 28
  Parental diary record of number of regurgitation per day reviewed at Day 0, Day 14 and Day 28

SECONDARY OUTCOMES:
Frequency of infant regurgitation | Day 0, Day 14, Day 28, and Age 8, 12, 16, 20 and 24 weeks
  Rome IV criteria diagnosed by physician
Frequency of infant colic | Day 0, Day 14, Day 28, and Age 8, 12, 16, 20 and 24 weeks
  Rome IV criteria diagnosed by physician
Frequency of functional constipation | Day 0, Day 14, Day 28, and Age 8, 12, 16, 20 and 24 weeks
  Rome IV criteria diagnosed by physician
Stool consistency | Day 0, Day 14, Day 28, and Age 8, 12, 16, 20 and 24 weeks
  Stool consistency based on Brussels infants and toddler stool scale (BITSS)
Stool frequency | Day 0, Day 14, Day 28, and Age 8, 12, 16, 20 and 24 weeks
  Number of defecations per day
Feeding difficulties | Day 0, Day 14, Day 28, and Age 8, 16 and 24 weeks
  NeoEAT questionnaire
Sleep | Day 0, Day 28, and Age 12 and 24 weeks
  Brief Infant Sleep questionnaire
Biochemical and metabolic markers: saliva markers | Day 0 and Day 14
  Saliva: inflammation markers (including enzymes reported in U/mL)
Biochemical and metabolic markers: saliva markers | Day 0 and Day 14
  Saliva: stress markers (including hormones reported in ng/mL)
Biochemical and metabolic markers: saliva markers | Day 0 and Day 14
  Saliva: inflammation markers (including proteins reported in µg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Sirinuch Chomtho, MD, PhD, Principal Investigator — Chulalongkorn University
Locations (1):
- Pediatric Nutrition Research Unit, Faculty of Medicine, Chulalongkorn University and King Chulalongkorn Memorial Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided